CLINICAL TRIAL: NCT00501579
Title: Study of Difluprednate in the Treatment of Uveitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Responsible Party: Chief Medical Officer, Sirion Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ST-601A-001
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — difluprednate; prednisolone acetate

INTERVENTIONS:
Drug: Difluprednate
Drug: Prednisolone Acetate

SUMMARY:
The purpose of this study is to determine the safety and efficacy of difluprednate compared with prednisolone acetate in the treatment of endogenous anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endogenous anterior uveitis in at least 1 eye

Exclusion Criteria:

* Presence of intermediate uveitis, posterior uveitis or panuveitis
* Corneal abrasion
* Any confirmed or suspected active viral, bacterial, or fungal keratoconjunctival disease
* Allergy to similar drugs, such as other corticosteroids

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Chair — Sirion Therapeutics
Locations (1):
- John-Kenyon American Eye Institute, New Albany, Indiana, United States

REFERENCES:
- [Derived] Foster CS, Davanzo R, Flynn TE, McLeod K, Vogel R, Crockett RS. Durezol (Difluprednate Ophthalmic Emulsion 0.05%) compared with Pred Forte 1% ophthalmic suspension in the treatment of endogenous anterior uveitis. J Ocul Pharmacol Ther. 2010 Oct;26(5):475-83. doi: 10.1089/jop.2010.0059. PMID 20809807